CLINICAL TRIAL: NCT03258775
Title: Water Consumption, Hydration and Resting Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 750014-4
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Hydration and Resting Metabolism
Keywords: RMR; hydration; substrate oxidation
MeSH Terms: interventions — Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 250ml (Active Comparator)
  Interventions: Other: water intake
- 500ml (Active Comparator)
  Interventions: Other: water intake

INTERVENTIONS:
Other: water intake — After an overnight fast participants' RMR will be measured by indirect calorimetry for 30 minutes after which either a low (250ml) or high (500ml) dose of water will be consumed followed by an additional 90 minutes of indirect calorimetry. The test day will be repeated after 7-10 days with the second dose of water. The order in which the dose of water will be consumed will be randomized

SUMMARY:
A randomized, cross over study will assess the effects of ingestion of high and low volumes of water on REE over 90 minutes. The high volume of water 500ml and the low volume of water 250ml. Participants will be computer randomized to determine which volume of water to receive first. Participants will arrive at the Nutrition Assessment Laboratory between 7:00 and 7:30am following a 9 hour overnight fast. Participants will be instructed not to consume any food or drink after 10pm the night before the assessment. Participants will also be asked to abstain from alcohol and caffeine for 3 days before the assessment. After verification of eligibility, baseline REE will be measured for 30 minutes followed by administration of first assigned dose of water. REE will be monitored for the next 90 minutes. Blood pressure and heart rate will also be monitored, simultaneously to REE. After a 7-10 day washout period, participants will return for their second test day where the second dose of water will be administered. A 7-10 day washout period was selected to allow participants time to resume normal diet and hydration between visits.

ELIGIBILITY:
Inclusion Criteria:

* 18-39 years of age
* Generally Healthy men and women
* BMI 18.5-28
* Willing to abstain from caffeine for 3 days prior to testing
* Able to provide written consent in English
* Ability to communicate in English (oral and written

Exclusion Criteria:

* <18 or >39 years
* BMI < 18.5 or >28
* Pregnant or Nursing
* Taking prescribed or over the counter medication affecting fluid balance or metabolism
* Suffers from hepatic, renal, pulmonary, endocrine or hematological disease
* Performs more than 3 hours a week of strenuous exercise
* Consumes, on average, more than 2 alcoholic beverages per day
* More than 5kg of weight change over the past 6 months
* Claustrophobic

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Resting Metabolic Rate (RMR) | 90 minutes
  Resting Metabolic Rate after water intake
Substrate oxidation | 90 minutes
  Change in substrate oxidation after water intake

SECONDARY OUTCOMES:
blood pressure | 90 minutes
heart rate | 90 minutes

IPD SHARING:
Plan to Share IPD: No